CLINICAL TRIAL: NCT00214825
Title: Aldosterone and Vascular Disease in Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Gail K. Adler, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-001273 BWH
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus; Endothelial Dysfunction; Albuminuria
MeSH Terms: conditions — Diabetes Mellitus; Albuminuria | interventions — Eplerenone; Hydrochlorothiazide

ARMS (2):
- 1 (Experimental): MR antagonist (Eplerenone) + placebo
  Interventions: Drug: eplerenone
- 2 (Placebo Comparator): Hydrochlorothiazide plus potassium
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: eplerenone — 50 mg daily for 6 weeks with placebo
  Arms: 1
Drug: Hydrochlorothiazide — HCTZ 12.5 mg with potassium (10 mEq) daily for 6 weeks
  Arms: 2

SUMMARY:
Specific aims for this proposal are to determine in patients with diabetes mellitus the effects of an aldosterone receptor antagonist on:

1. Coronary microvascular function assessed by MRI perfusion reserve,
2. Endothelial dysfunction assessed by brachial artery reactivity studies, and
3. Inflammation assessed by blood measurements of c-reactive protein (CRP), monocyte chemoattractant protein-1 (MCP-1), and plasminogen activator inhibitor-1 (PAI-1).

DETAILED DESCRIPTION:
Recent human and animal studies suggest that activation of the mineralocorticoid receptor (MR) by aldosterone, the final product of the renin-angiotensin-aldosterone system, causes microvascular damage, vascular inflammation, and endothelial dysfunction. Angiotensin converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBs) are unable to provide long-term aldosterone suppression. Therefore, we hypothesize that activation of the MR contributes to progression of vascular disease in patients with diabetes already using ACE inhibitor therapy.

Specific aims for this proposal are to determine in patients with type 1 or type 2 diabetes mellitus and proteinuria, already receiving ACE inhibitor or ARB therapy, the effects of an aldosterone receptor antagonist vs. hydrochlorothiazide on:

1. Coronary microvascular function assessed by MRI perfusion reserve,
2. Endothelial dysfunction assessed by brachial artery reactivity studies,
3. Inflammation and cellular oxidative stress and injury, assessed by c-reactive protein (CRP), MCP-1, plasminogen activator inhibitor-1 (PAI-1).
4. Proteinuria and whether there is a differential effect when a MR antagonist or HCTZ is added to the ACE inhibitor therapy.

This is a double-blind, randomized, cross-over study of men and women (21-64 years old) with type 1 or type 2 diabetes mellitus and albuminuria (³30 mg/g creatinine). Participants will be randomized to a MR antagonist + placebo or HCTZ + potassium supplementation for 6 weeks. The MR antagonist arm will receive eplerenone 50 mg daily. The HCTZ arm will receive HCTZ 12.5 mg with potassium 10 Meq daily. Amlodipine 5 to 10 mg daily will be added during run phase to control blood pressure. Blood pressure goal is less than 130/80 mm Hg. There will be a 4-week washout period before the patients are crossed-over to the other study arm. MRI perfusion reserve, brachial artery reactivity, and blood samples will be obtained at the beginning and end of each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

Men and women (21-64 years old) with type 1 or type 2 diabetes mellitus and albuminuria (over 30 mg/g creatinine).

Exclusion Criteria:

Exclusion criteria include: (1) subjects without hypertension who have baseline systolic blood pressure <100 mmHg, (2) severe hypertension (blood pressure must be well-controlled on 3 antihypertensive agents or <150/100 mmHg on £2 antihypertensive agents), (3) ischemic changes on resting electrocardiogram, (4) clinical evidence of heart disease, cerebrovascular or peripheral vascular disease, (5) significant cardiac arrhythmias, (6) aortic stenosis, (7) 2nd or 3rd degree atrio-ventricular block, sinus node disease, or symptomatic bradycardia, (8) bronchospastic lung disease with active wheezing, (9) known hypersensitivity to any of the study drugs, (10) any contraindication to MRI, (11) serum creatinine ³ 1.5 mg/dL, (12) serum potassium ³ 5.0 mmol/L, (13) current smoker, (14) Serum transaminases greater than twice the upper limit of normal, (15) a history of gout, (16) pregnancy, and (17) other active medical problems detected by examination or laboratory testing.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2003-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Coronary microvascular function assessed by myocardial perfusion reserve measured by MRI | 20 weeks

SECONDARY OUTCOMES:
Endothelial dysfunction assessed by brachial artery reactivity | 20 weeks
Inflammation and cellular oxidative stress and injury, assessed by CRP, MCP-1, PAI-1, nephrin, cystanin C, F2 isoprostanes, and urinary 12-HETE | 20 weeks
Proteinuria | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital Boston, MA
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Joffe HV, Kwong RY, Gerhard-Herman MD, Rice C, Feldman K, Adler GK. Beneficial effects of eplerenone versus hydrochlorothiazide on coronary circulatory function in patients with diabetes mellitus. J Clin Endocrinol Metab. 2007 Jul;92(7):2552-8. doi: 10.1210/jc.2007-0393. Epub 2007 May 8. PMID 17488800